CLINICAL TRIAL: NCT06575283
Title: Early Prediction of Cerebral Palsy by MRI in Infants With White Matter Injury: a Multicenter Study
Brief Title: Predicting Cerebral Palsy in Infants With White Matter Injury Using MRI
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Shenzhen Children's Hospital (Other Government); Zunyi Medical College (Other); Wuxi Women's & Children's Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Chengdu Medical College (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Baoji Central Hospital (Other); Xian Children's Hospital (Other Government); Guangzhou Women and Children's Medical Center (Other); Third Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2024LSYY-154
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy; Periventricular White Matter Abnormalities
Keywords: Cerebral palsy; Periventricular white matter injury; MRI; Deep learning
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PVWMI Infants aged 6 months to 2 years: Infants will be scanned by MRI at the age of 6 months to 2 years. The infants of periventricular white matter injury (PVWMI) will be enrolled.
  Interventions: Other: No intervention will be performed in this cohort study

INTERVENTIONS:
Other: No intervention will be performed in this cohort study — Deep learning classification models will be used for automatic prediction of cerebral palsy. Machines will be used to assist doctors in cerebral palsy risk evaluation.

SUMMARY:
The goal of this study is to determin the MRI features associated with cerebral palsy and to develop prediction models of pediatric disorders by combining MRI with artificial intelligence.

The main questions it aims to answer are:

* How to achieve features on conventional MRI associated with cerebral palsy?
* How to predict the risk of cerebral palsy in infants aged 6 to 2 years based on conventional MRI and deep learning? Researchers will compare characteristics of periventricular white matter injury with cerebral palsy to those without cerebral palsy.

Participants will be asked to provide MRI data, clinical diagnoses information, and follow-up outcomes.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a common group of movement disorders that often results in disability in children. In the context of CP, the importance of early diagnosis is crucial, but current diagnostic modalities often identify cases after the age of 2 years. After initial screening of infants at high risk for CP by behavioral scoring, magnetic resonance imaging (MRI) forms an integral part of the comprehensive evaluation. The training of conventional model of CP risk prediction requires a large investment of time and financial resources. The average sensitivity rate drops to 90%. Up to now, deep learning technology has been widely used in tasks related to image-based disease classification and has shown excellent performance.

Periventricular white matter injury (PVWMI) accounts for the largest proportion of various types of brain injuries in cerebral palsy, and the types of brain injuries in cerebral palsy are rich and complex, posing difficulties and challenges to deep learning models. Therefore, this study focuses on PVWMI, the most common type of cerebral palsy, and uses conventional MRI to develop a deep learning prediction model for CP in infants aged 6 months to 2 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children at high risk of periventricular white matter injury (PVWMI) (gestational age <35 weeks, birth weight <2.6 kg, forceps-assisted delivery/fetal head attraction, Apgar score <7, hypoglycaemia, sepsis, electrolyte disturbances, premature rupture of membranes);
2. Those who underwent MRI at 6 months of age-2 years, including at least T1WI and T2WI sequences;
3. Upon follow-up, the patient's clinical diagnosis: cerebral palsy, other diagnoses that did not develop into cerebral palsy, or inability to confirm the diagnosis).

Exclusion Criteria:

1. Incomplete MRI images or unreadable images due to motion artefacts;
2. Incomplete neurobehavioural assessment data (including: gross motor function).

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will follow up infants from multiple regions and different hospitals who underwent MRI examinations between 6 months and 2 years old. Each infant and young child included T1-weighted imaging (T1WI) and T2-weighted imaging (T2WI). According to the follow-up outcomes, these infants will be divided into the following groups: cerebral palsy, other diagnoses that did not develop into cerebral palsy, or inability to confirm the diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the model predicting cerebral palsy | From September 2024 to December 2025
  Determine the accuracy of PVWMI classification and cerebral palsy prediction. The higher the value, the better the model performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, Ph.D.,M.D, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after the paper published.
Access Criteria: The data can be used just for research purpose. Users can contact to the corresponding author through e-mail.